CLINICAL TRIAL: NCT00797615
Title: Project Diabetes: Weight Gain Prevention in Hispanic Girls (GEMAS Study)
Acronym: GEMAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Bettina M. Beech, DrPH, MPH, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 081057
Record Dates: First submitted 2008-11-21; First posted 2008-11-25 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2010-10

CONDITIONS: Obesity; Diet; Exercise; Behavioral Research
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alternative Intervention (Placebo Comparator): 12-week alternate intervention program focused on building self-esteem and social self-efficacy
  Interventions: Behavioral: Alternative Intervention
- Active Intervention (Active Comparator): 12-week intervention program focused on dietary intake and physical activity
  Interventions: Behavioral: Active intervention

INTERVENTIONS:
Behavioral: Active intervention — 12-week family-based weight gain intervention program focused on dietary intake and physical activity for 8-10 year old Hispanic girls and their parents (N=30 girl-parent dyads).
  Arms: Active Intervention
Behavioral: Alternative Intervention — 12-week alternative intervention addressing self-esteem, for 8-10 year old Hispanic girls and their parents (N=30 girl-parent dyads).
  Arms: Alternative Intervention

SUMMARY:
Over the past 30 years obesity has reached epidemic proportions in the United States (Ogden et al, 2006). While this epidemic affects all socioeconomic levels, certain racial/ethnic groups such as Hispanics, are disproportionately affected by obesity and diabetes. The age of onset of excess obesity in Hispanic females, formerly young adulthood, is now younger. Childhood obesity poses intermediate and long-term health risks, including: type 2 diabetes, hyperlipidemia, elevated blood pressure, and metabolic syndrome. Although biological factors may influence a child's risk for becoming overweight, the home environment has been shown to be a predisposing and reinforcing contextual factor for unhealthy eating and exercise behaviors. Since parents are the primary transmitters of Hispanic cultural practices and significantly influence their children's diet and physical activity behaviors from preschool through high school, family-based weight-gain prevention interventions are likely to be effective.

The goal of this implementation study is to contribute to the reduction of racial/ethnic disparities in obesity and risk of type 2 diabetes by tailoring a recently successful childhood obesity prevention program originally developed for African American girls to implement and evaluate with preadolescent Hispanic girls.

DETAILED DESCRIPTION:
Over the past 30 years obesity has reached epidemic proportions in the United States (Ogden et al, 2006). While this epidemic affects all socioeconomic levels, certain racial/ethnic groups such as Hispanics, are disproportionately affected by obesity and diabetes. The age of onset of excess obesity in Hispanic females, formerly young adulthood, is now younger. Childhood obesity poses intermediate and long-term health risks, including: type 2 diabetes, hyperlipidemia, elevated blood pressure, and metabolic syndrome (Goran et al 2003; Hale and Rupert, 2006). Although biological factors may influence a child's risk for becoming overweight, the home environment has been shown to be a predisposing and reinforcing contextual factor for unhealthy eating and exercise behaviors (Arredondo et al, 2006).

Two recent empirical reviews of childhood obesity interventions demonstrated the increased effectiveness of family-based approaches (Kitzmann and Beech, 2006; Summerbell et al, 2007). Since parents are the primary transmitters of Hispanic cultural practices and significantly influence their children's diet and physical activity behaviors from preschool through high school (Snethen et al, 2007), family-based weight-gain prevention interventions are likely to be effective. The sociocultural context of Hispanic girls involves a much higher degree of interdependence among family members in Hispanic compared to White families (Schwartz, 2007). In addition to family-based approaches to pediatric obesity prevention, culturally-relevant and community-based participatory approaches have been strongly recommended by the Institute of Medicine (IOM) and the Strategic Plan for NIH Obesity Research (NIH, 2004:25).

The goal of this implementation study is to contribute to the reduction of racial/ethnic disparities in obesity and risk of type 2 diabetes by tailoring a recently successful childhood obesity prevention program originally developed for African American girls to implement and evaluate with preadolescence Hispanic girls. This project will be a collaborative, participatory community-academic partnership between Vanderbilt University Medical Center (VUMC), Tennessee State University (TSU) Center for Health Research, Meharry Medical College, Progreso Community Center (PCC) and the Nashville Latino Health Coalition (NLHC). Specifically, the childhood obesity prevention program called Girl's health Enrichment Multi-site Studies (GEMS) will be tailored to be culturally-appropriate and piloted in the Hispanic/Latino community in Nashville/Davidson County, Tennessee. Dr. Bettina Beech led the development of the original GEMS intervention, which was developed and pilot-tested in Memphis, Tennessee (Beech et al, 2003). We have assembled a multi-disciplinary team with expertise in pediatric obesity (Drs. Beech, Barkin, and Cook), type 2 diabetes (Dr. Tom Elasy), community-based participatory research (Drs. Beech, Barkin, Hull), Hispanic culture (Drs. Hull and Zoorob, PCC), and community engagement (NLHC, PCC, and Drs. Beech and Hull).

ELIGIBILITY:
Inclusion Criteria:

* 8-10 year old Hispanic girls in Nashville
* The parent or guardian must identify the girl as Hispanic
* The parent or guardian must identify that the girl be at or above the 25th percentile of age- and sex-specific BMI based on the 2000 CDC growth charts or one parent/caregiver must have BMI>25 kg/m2.

Exclusion Criteria:

* Baseline girls' BMI>35
* Medical conditions and medications affecting growth
* Conditions limiting participation in the interventions (e.g., unable to participate in routine physical education classes in school)
* Conditions limiting participation in the assessments (e.g., two or more grades behind in school for reading and writing)
* Other criteria (e.g., inability or failure to provide informed consent).

Ages: 8 Years to 10 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 132 (Actual)
Dates: Start 2008-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the between-group differences in BMI and body fat. | After 12 weeks of intervention

SECONDARY OUTCOMES:
Secondary outcomes will include dietary intake and physical activity. | After 12 weeks of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Bettina M. Beech, DrPH, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (2):
- United States (2):
  - Progreso Community Center, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee